CLINICAL TRIAL: NCT01241370
Title: Skin and Retina Microvascular Endothelial Function in Healthy, Insulin Resistant and Type 2 Diabetic Subjects
Status: Completed | Type: Observational
Sponsor: ELAB-Logistics (Industry)
Collaborators: Institute for Clinical Research and Development (ikfe) GmbH (Unknown); Johannes Gutenberg University Mainz (Other); University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Prof. Dr. Thomas Forst / CEO ikfe GmbH, ikfe GmbH
Other Study IDs: IKFE-RET-001
Record Dates: First submitted 2010-11-10; First posted 2010-11-16 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Retinal endothelia dysfunction; Type 2 diabetes mellitus; Insulin-resistance; micro-lightguide spectrophotometry; laserdopplerfluxmetry
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Lean healthy subjects: Homeostasis Model Assessment score (HOMAs) ≤ 2, Body Mass Index (BMI) ≤ 28 kg/m2
- Insulin-resistnat subjects: HOMAs > 2, BMI > 28 kg/m2
- Type 2 diabetic patients

SUMMARY:
The purpose of this study is to investigate microvascular endothelial function in the retina of lean, obese, and type 2 diabetic subjects and to compare microvascular endothelial function in the retina with several other established markers of endothelial and microvascular function.

DETAILED DESCRIPTION:
Insulin resistance is an early feature in obese patients lasting from hyperinsulinaemia with normal glycaemic control to impaired glucose tolerance and clinically manifest type 2 diabetes. Insulin resistance is closely associated to endothelial dysfunction and many other cardiovascular risk markers summarised under the definition of the metabolic syndrome. During the recent years, insulin resistance and the development of endothelial dysfunction were recognized as important pathogenetic drivers in the development of atherosclerosis and major predictors in the development of micro and macrovascular complications like retinopathy, nephropathy, myocardial infarction or stroke.

Several different technologies have been developed for the measurement of endothelial function in distinct vascular compartments like the flow mediated vasodilatation in the brachial artery, or numerous laser Doppler based technologies for the measurement of endothelial dependent microvascular blood flow responses in the skin. Even retinal vascular morphology could be easily visualized by direct fundoscopy, the investigation of retinal endothelial function had been a diagnostical challenge for decades. During the recent years, laser doppler scanning of the retina has become a widely used technology for the measurement of microvascular blood flow in the retina. Recently a new stimulation technology for the investigation of endothelial function in the retina has been developed and validated. Application of flickering light to the retina increases retinal blood flow by the stimulation of endothelial nitric oxide (NO) release, and laser Doppler scanning of the retina before and after the flicker light application could be used for the investigation of microvascular endothelial function in the eye. For assessing the stage of retinopathy a retinal image of 45° (papilla-centered) will be performed using a digital non-mydriatic fundus camera (Kowa Nonmyd 5). The image will be evaluated in respect to diabetic and hypertensive retinopathy in a standardized method. Also the equivalent arteriolar and venous diameter of the retinal vessels will be measured and the arterio-venous ratio will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age: 30 to 70 years
* Have given informed consent to participate in this study in accordance with local regulations
* Are reliable and willing to make themselves available for the duration of the study and will abide by the study restrictions

Exclusion Criteria:

* Smoking within the last 6 months
* Pre-proliferative or proliferative diabetic retinopathy
* Have a history of drug or alcohol abuse within the last 5 years
* Pregnant or intend to become pregnant during the course of the study
* Have a condition (including known drug abuse, alcohol abuse, or psychiatric disorder) which, in the opinion of the investigator, precludes the patient from following and completing the protocol
* Epilepsy
* Lack of compliance or another, similar reason, that, in the judge of the investigator, precludes satisfactory participation in the study.
* Treatment with nitrates, angiotensin converting enzyme (ACE)-inhibitors, or angiotensin (AT) II blockers
* Treatment with glitazones

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is planned to recruit up to 60 obese male and female subjects, stratified according to the following,
  20 non-diabetic subjects with HOMAs ≤ 2, BMI < 28 kg/m² 20 non-diabetic subjects with HOMAs > 2, BMI ≥ 28 kg/m² 20 type 2 diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2009-05; Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Comparison of retinal microvascular endothelial function in obese insulin sensitive, insulin-resistant and type 2 diabetic subjects with retinal microvascular endothelial function in lean healthy control subjects. | 2-28 days
  Measurements were taken from the superficial retinal layer (300 µm) using a scanning laser doppler flowmetry at 720 nm (Heidelberg Retina Flowmeter, Heidelberg Engineering)

SECONDARY OUTCOMES:
Comparison of microvascular endothelial function in the skin in obese and type 2 diabetic subjects with microvascular endothelial function in lean healthy control subjects. | 2-28 days
  A simultaneous micro-lightguide spectrophotometry and laserdoppler-fluxmetry were used to measure the microvascular skin blood flow and postcapillary tissue oxygenation in a depth of 2 mm at the lower forearm (oxygen to see (O2C), Lea Medizintechnik, Giessen, Germany).
Comparison of microvascular endothelial function in the retina with microvascular endothelial function in the skin in diabetic and in non-diabetic subjects. | 2-28 days
Comparison of morphologic changes in retinal vessels (atrio-venous-ratio, diameter) in diabetic and in non-diabetic subjects. | 2-28 days
Comparison of the Oral Glucose Tolerance Test (OGTT) in the different subject groups with skin and retinal endothelial function. | 2-28 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Forst, MD, Principal Investigator — Ikfe GmbH
Locations (1):
- ikfe GmbH, clinic, Mainz, Germany